CLINICAL TRIAL: NCT00160888
Title: Endothelium-Dependent Vasoreactivity in Nitric Oxide Synthase Gene (Glu298Asp) Polymorphism: Studies in Healthy Volunteers
Brief Title: Vasoreactivity in Carriers of Genetic Polymorphisms
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: K004
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Healthy
MeSH Terms: interventions — Nitroprusside; Bradykinin; Acetylcholine

INTERVENTIONS:
Drug: sodium nitroprusside, bradykinin, acetylcholine

SUMMARY:
The objective of the study is to assess the impact of genetic variation (especially polymorphisms of the gene coding endothelial nitric oxide synthase (eNOS) and the bradykinin B2 receptor gene) on venous and arterial responsiveness to vasodilators in healthy individuals without cardiovascular risk factors.

DETAILED DESCRIPTION:
Study I: Using the dorsal hand vein compliance technique dose-response curves to bradykinin and sodium nitroprusside will be obtained in healthy volunteers during preconstriction with phenylephrine and after pretreatment with a single dose of 500 mg i.v. acetylsalicylic acid.

Study II: Using venous occlusion plethysmography dose-response curves to acetylcholine, sodium nitroprusside and L-NG-monomethyl-arginine (L-NMMA) will be obtained in healthy volunteers pretreated with a single dose of 500mg i.v. acetylsalicylic acid.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 70
* gender: male
* good state of health

Exclusion Criteria:

* known condition causing endothelial dysfunction (e.g. diabetes, hyperlipidaemia, arterial hypertension, smoking, homocysteinemia)
* regular medication and/or treatment with drugs within the last 4-6 weeks (exclusion has to be decided in each case)
* acute or chronic illness
* methylxanthines and alcohol during 12 hours before the study
* nicotine during 1 year before the study
* drug and/or alcohol abuse
* pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1999-11; Study Completion 2006-12

PRIMARY OUTCOMES:
Study I: Venous responsiveness assessed by dorsal hand vein compliance technique
Study II: Forearm blood flow assessed by venous occlusion plethysmography

CONTACTS AND LOCATIONS:
Overall Officials: Walter E Haefeli, MD, Principal Investigator — Dept. of Internal Medicine VI, University of Heidelberg
Locations (1):
- Dept. of Internal Medicine VI, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Fricker R, Hesse C, Weiss J, Tayrouz Y, Hoffmann MM, Unnebrink K, Mansmann U, Haefeli WE. Endothelial venodilator response in carriers of genetic polymorphisms involved in NO synthesis and degradation. Br J Clin Pharmacol. 2004 Aug;58(2):169-77. doi: 10.1111/j.1365-2125.2004.02130.x. PMID 15255799